CLINICAL TRIAL: NCT02941770
Title: The Effect of a Physical Activity Consultation in the Management of Adolescent Overweight, Including Anthropometry, Physical Activity Levels, Cardiorespiratory Fitness, and Endothelial Health
Brief Title: Physical Activity Consultation in the Management of Adolescent Overweight
Acronym: PAC-MAnO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, A. Videira-Silva, PhD student, University of Lisbon
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1332/CC1942016
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Overweight
Keywords: Adolescents; Overweight; Obesity; Weight Loss; Physical activity consultation; Cardiorespiratory fitness; Endothelial structure; Endothelial function
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Clinic standard care protocol:
  * Baseline evaluation session with a Pediatrician for initial screening;
  * Appointment with a Dietitian;
  * A brochure with physical activity guidelines for youth with examples of physical exercises.
- Intervention group I (Experimental): * Clinic standard care protocol;
  * Physical activity consultation (Physical activity behavior change);
  Interventions: Behavioral: Physical activity behavior change
- Intervention group II (Experimental): * Clinic standard care protocol;
  * Physical activity consultation;
  * 2 exercise sessions per week (≈60 min/session) directed by one Exercise Physiologist.
  Interventions: Behavioral: Physical activity behavior change; Other: Exercise

INTERVENTIONS:
Behavioral: Physical activity behavior change — Physical activity consultation will consist in a patient-centered, one-to-one session based on the transtheoretical model and will use motivational interview in order to strengthen individual's intrinsic motivation to achieve a positive PA behavior change. In these sessions the following topics will be explored: (i) explore and resolve ambivalence; (ii) identify difficulties/barriers, and benefits of behavior change; (iii) find their own means and their own solutions for step over the identified barriers; (iv) enhancement of autonomy and self-efficacy.
  Arms: Intervention group I; Intervention group II
Other: Exercise — Experimental group II will participate accordingly with their availability in two exercise sessions per week (≈60 min/session) directed by one exercise physiologist. The ability to exercise will be assessed in order to customize the exercise plan. All the sessions will include: 10 minutes of warm-up, 5 minutes of agility exercises, 15 minutes of resistance training (including the major upper and lower muscles, 12-15 sets of 15 repetitions), 20 minutes of aerobic exercise, and 10 minutes of cool-down (50-80% heart rate reserve - Polar Vantage NV, Polar Electro Oy, Kempele, Finland). All the participants will have to attend at least 80% of the scheduled sessions.
  Arms: Intervention group II

SUMMARY:
The prevalence of pediatric obesity makes this condition a worldwide public health concern. Physical Activity (PA) is recognized as having many health benefits, many of them related to obesity and its comorbidities. Despite of all the efforts, the majority of the overweight children/adolescents still present low levels of PA and high levels of sedentary behaviors. Thus, it seems that the greatest challenge is to influence behavior change in order to increase PA exposure in this population. PA consultation can be a cost-effective way of enhancing PA and improve weight status among overweight children.

The main objective of this study is to analyze if the inclusion of a PA consultation in a multidisciplinary program for the management of adolescent overweight improves body mass index (BMI) z-score, PA levels and sedentary behavior outcomes at six and twelve months, compared to those attending only the Pediatric and the Dietetic consultations.

This study was designed as a non-randomized, controlled clinical trial with six months duration and follow-up at the 12th month, that will include overweight adolescents (BMI ≥ p85) aged 12 to 17, attending the Clinic for the first time, and accepted to be enrolled. Those with (i) major pathologies (other than obesity or its related comorbidities), (ii) inability to perform regular PA, (iii) mental disorders, (iv) smoking habits, (v) under any kind of prescription (other than antihypertensives or metformin), or (vi) being involved in another weight loss program will be excluded. According to the sample size calculation, we expect to recruit 129 participants that will be allocated in three groups by consecutive sampling: (i) control group - standard care (Pediatric and Dietitian consultations); (ii) intervention group I - standard care plus PA consultation; (iii) intervention group II - 2 weekly exercise sessions additionally to the standard care and PA consultations..

DETAILED DESCRIPTION:
Secondary objectives

The success of adolescent obesity management cannot be assessed only based on the BMI/BMI z-score or PA levels. Thus, the secondary objectives of this study are:

(i) Analyze the effect of the intervention on cardiorespiratory fitness (CRF). CRF is commonly expressed as VO2 max and represents the ability to uptake, deliver, and use oxygen to produce energy. CRF is inversely associated with BMI and waist circumference, and have a potential beneficial effect on the endothelial function and structure - which is known to be impaired among overweight adolescents - even without the occurrence of major changes in the BMI.

(ii) Analyze the effect of the intervention on biochemical markers, including insulin resistance and lipid profile.

(iii) Analyze whether changes in BMI z-score, PA/sedentary behavior and CRF are associated with changes in endothelial structural health (assessed trough carotid intima-media thickness - cIMT) and function (assessed trough pulse wave velocity - PWV).

(iv) Validate a sub-maximal exercise step test for an overweight adolescent population for future use in the PA consultation routine. Sub-maximal exercise step testing has been considered a timely and cost-effective method of assessing CRF, which can be conducted at the clinical office with minimal risk and discomfort for the participant compared to maximal exercise testing.

(v) Analyze the cost-effectiveness (CE) of the intervention, since it is considered as an important aid to public health decision-making, with an extra potential additional value in a tertiary health care setting.

Data collection methods

Socio-economic status Social-economic classification (SES) will be based on the parents/caregivers occupation, according to the Portuguese National Institute of Statistics. The socio-occupational status of both parents/caregivers will be categorized in three groups: (i) management positions (Class I); (ii) office, service or skilled manual workers (Class II and III); (iii) unskilled workers or unemployed (Classe IV and V).

Anthropometry The anthropometric assessments will be performed at the exercise physiologist office in the outpatient clinic, Department of Pediatrics, HSM. All the assessments will be performed by the same investigator. With the exception of body composition, all the other anthropometric assessments will be performed twice as a confirmation procedure. The Technical Error of Measurement (TEM) will be calculated accordingly to: TEM=√[∑Dif2/2n]).

(i) Height (height stadiometer, SECA 217, Hamburg, Germany) assessed in the anthropometric position, without shoes, with the participant back to the stadiometer, and after an expiratory phase. Height will be registered to the nearest 0.1 cm; (ii) Body weight and body composition (bioelectrical impedance scale InBody 230, Seoul, Korea). Body weight will be measured to the nearest 0.1 kg, in the anthropometric position (with the palms turned into thighs), with the subjects wearing as few clothes as possible, and without shoes or socks; (iii) BMI will be calculated as body weight in kilograms divided by the square of height in meters [BMI= weight (kg)/height2 (m)]. We will further calculate the BMI z-score [BMI z-score= [(BMI/M(t))L(t)-1]/L(t)S(t)], since it is acknowledge as the best choice to track changes in growing children; (iv) Waist and hip circumferences (circumference measuring tape, SECA 203, Hamburg, Germany) will be measured with the subject standing. Waist circumference will be measured 1 cm above the iliac crest at the end of a regular expiration, and hip circumference at the maximum protuberance of the buttocks.

Body Composition (Dual-energy X-ray absorptiometry) Additionally to bioelectrical impedance, which is a usual assessment in the clinical office, body composition will be assessed by DXA (Explorer W, Hologic; Waltham, MA, USA) and analyzed using the equipment's software (QDR 12.4, Waltham, MA, USA). DXA exam will be performed in accordance with the National Health and Nutrition Examination Survey (NHANES) protocol. Trunk and Whole Body Fat, as well as Trunk and Whole Body Peripheral Fat will be assessed. All the procedures will be performed by the same investigator. All the scans will be made in the morning after overnight feasting (10-12 hours).

Clinical assessments (i) Pubertal status will be assessed by a pediatrician and categorized in accordance with Tanner stages.

(ii) Resting blood pressure (digital sphygmomanometer, CAS 9302S, CAS Medical Systems, Branford, USA) will be measured in the right arm with an appropriate sized cuff, after five minutes of rest in the seating position. The measurement will be performed three times and the average of the three measurements will be recorded. Children will be then classified accordingly to sex, age and height-specific charts.

(iii) Biochemical analysis will be performed in the laboratory of clinical pathology at the HSM. Blood samples will be collected after overnight feasting (10-12 hours) in the presence of one of the parents/ caregivers, and after a local application of a topical anesthesia patch (EMLA). Blood glucose levels will be determined using hexokinase method and insulin will be assessed using a chemiluminescence immunoassay technique. Insulin sensitivity will be derived from the homeostasis model assessment (HOMA) method. Total cholesterol, triglycerides, and high density lipoprotein cholesterol will be determined using enzymatic, GPO-trinder, and direct methods, respectively. Plasma liver enzymes (AST, ALT, and GGT) will be assessed with modified IFCC method. C-reactive protein will be determined using a turbidimetric immunoassay (Siemens, ADVIA 2400, Newark, DE, USA).

Energy intake A three-day food record (2 weekdays and 1 weekend day) using semi-quantitative scaling (e.g. number of spoons or scoops) will be used in order to provide comprehensive information about meal patterns and to estimate the energy intake. Although it is known that overweight children tend to underestimate their energy intake, the 3-day food diary still is considered acceptable and often used instrument at the clinical practice. Moreover, the use of a 3-day food diary instead of a 7-day, may enhance the adherence to the instrument.

Physical activity, sedentary behaviors and cardiorespiratory fitness Data from the accelerometers will be uploaded at the Exercise and Health Laboratory, Faculty of Human Kinetics, University of Lisbon, Lisbon, Portugal. Sedentary activity questionnaires and CRF will be assessed at the same institution.

(i) PA will be assessed with accelerometers (ACTIGRAPH GT3X, Pensacola, Florida, USA). All the subjects will use one accelerometer above the right hip, near to the iliac crest, during at least one weekend day and two week days, except during sleep, bath or swimming. The accelerometer will be programmed to use a 5-second cycle. Only days with more than 480 min (8h) counted, will be considered into the analysis. Periods of 60 min with "zero activity" will be interpreted as un-using equipment. The data upload will be performed with the ActiLife software, version 6.8.0. Between 0 and 149 counts/minute we will consider as sedentary activity; between 150 and 499, Light Physical Activity (LPA); between 500 and 3999, Moderate Physical Activity (MPA); between 4000 and 7599, Vigorous Physical Activity (VPA); and with more than 7600 counts/minute Very Vigorous Physical Activity (VVPA); (ii) Sedentary behaviors will be assessed by a questionnaire (questionnaire ASAQ - adolescent sedentary activity questionnaire) additionally to the accelerometry, answered while waiting for the assessment of CRF. The ASAQ is a reliable and cost-effective instrument that may be able to measure three dimensions of the sedentary behaviors (type, frequency and time/duration).

(iii) CRF will be indirectly determined with a maximal exercise test using a cycle ergometer (electronically braked cycle ergometer, Monark 839 Ergomedic, Monark, Vansbro, Sweden). Initial workload and increments will be of 40 or 50 W for girls and boys, respectively. Heart rate will be registered continuously (Polar Vantage NV, Polar Electro Oy, Kempele, Finland). Criteria to stop the test will include a heart rate superior to the theoretical maximal heart rate (208 - 0.7(age), failure to maintain a frequency of at least 30 revolutions/min, and a subjective judgement by the observer that the adolescent is exhausted. The maximal power output (Wmax) will be calculated as the power in the last fully completed workload plus the power increment of the last step multiplied by the time proportion completed of the last step. The maximal power output will be converted to VO2 (ml/kg/min) using the following equation: VO2 (1∕min) = 0.465 + (0.0112 ×Wmax) + (0.172 × sex), where sex =0 for girls and sex=1 for boys (38).

Carotid intima-media thickness and pulse wave velocity cIMT and pulse wave velocity will be measured in the Exercise and Health Laboratory, Faculty of Human Kinetics, University of Lisbon, Lisbon, Portugal.

(i) cIMT will be measured with an ultrasound imager using a 13 MHz probe (MyLab One, Esaote, Genoa, Italy). cIMT will be defined as the distance between the lumen-intima and the media-adventitia interfaces. The measurement will be performed in the longitudinal plane on the right carotid artery, accordingly with previously validated radiofrequency-based tracking of arterial wall that allows a real-time determination of common carotid far-wall thickness (QIMT®) with high spatial and temporal resolution. cIMT will be automatically measured, and distension curves will be acquired within a CCA 1.59-cm region of interest, approximately 1 cm proximal to the carotid bifurcation. Maximum and minimum carotid diameters will be obtained from the distension curves.

(ii) PWV will be measured with applanation tonometry immediately after ultrasound imaging. Pressure curves from left carotid, femoral, radial and distal posterial tibial arteries will be assessed with two specific pressure sensitive transducers. The distance between the carotid and femoral, radial and distal posterial tibial arteries, will be measured directly and entered into the Complior Analyse software (ALAM Medical, Paris, France). Left brachial blood pressure will be measured and entered into the software. The values obtained from the carotid to femoral artery (aortic), carotid to radial artery (upper limb) and carotid to distal posterior tibial artery (lower limb) will be recorded as indices of central/aortic, upper and lower limb arterial stiffness, respectively.

Statistical methods Statistical analysis will be performed using the software IBM SPSS statistics (IBM SPSS statistics, version 22.0, IBM, New York, USA). We intend to use the Chi-square and one-way analysis of variance (ANOVA) to evaluate baseline differences between the control and intervention groups. The effect of the intervention will be analyzed with analysis of co-variance (ANCOVA) controlling for baseline values of continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Coming from the Lisbon region;
* A BMI ≥ p85 for gender and age;
* Attending the Clinic for the first time;
* Accepted to be enrolled.

Exclusion Criteria:

* Major pathologies (other than obesity or its related comorbidities);
* Inability to perform regular PA;
* Mental disorders;
* Smoking habits;
* Under any kind of prescription (other than antihypertensives or metformin);
* Being involved in another weight loss program.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) z-score | 12 months
Physical activity (PA) levels | 12 months
Sedentary behavior | 12 months
  Questionnaire ASAQ (Adolescent Sedentary Activity Questionnaire)

SECONDARY OUTCOMES:
Cardiorespiratory fitness (CRF) | 12 months
  Maximal (Cycle ergometer and gas analyser) and submaximal (step) testes
Carotid intima-media thickness (cIMT) | 12 months
Pulse wave velocity (PWV) | 12 months
Body composition | 12 months
Lipid profile (TC, LDL-C, HDL-C) | 12 months
Glucose metabolism (Glucose, Insulin, HOMA-IR) | 12 months
inflammation (C-RP) | 12 months
Cost-effectiveness (CE) | 12 months
  CE will be estimated for the standard intervention, and for both the intervention groups. CE ratio = C/E, (where C = cost of each intervention [human and material resources in €]; and E = effectiveness of each intervention [BMI z-score outcome]. The lowest CE ratio will represent the most cost-effective intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Fonseca, MD, PhD, Study Director — Pediatric Obesity Clinic, Department of Pediatrics, Hospital de Santa Maria, Lisbon, Portugal
Locations (1):
- Hospital de Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCallum Z, Wake M, Gerner B, Baur LA, Gibbons K, Gold L, Gunn J, Harris C, Naughton G, Riess C, Sanci L, Sheehan J, Ukoumunne OC, Waters E. Outcome data from the LEAP (Live, Eat and Play) trial: a randomized controlled trial of a primary care intervention for childhood overweight/mild obesity. Int J Obes (Lond). 2007 Apr;31(4):630-6. doi: 10.1038/sj.ijo.0803509. Epub 2006 Dec 12. PMID 17160087
- [Background] Henderson M, Daneman D, Huot C, McGrath J, Lambert M, Hux J, Booth GL, Hanley A. The impact of exercise consultation on activity levels and metabolic markers in obese adolescents: a pilot study. Int J Pediatr Endocrinol. 2010;2010:681510. doi: 10.1155/2010/681510. Epub 2010 Sep 26. PMID 20976257
- [Background] Kelishadi R, Malekahmadi M, Hashemipour M, Soghrati M, Soghrati M, Mirmoghtadaee P, Ghatrehsamani S, Poursafa P, Khavarian N. Can a trial of motivational lifestyle counseling be effective for controlling childhood obesity and the associated cardiometabolic risk factors? Pediatr Neonatol. 2012 Apr;53(2):90-7. doi: 10.1016/j.pedneo.2012.01.005. Epub 2012 Mar 3. PMID 22503255
- [Background] Walpole B, Dettmer E, Morrongiello BA, McCrindle BW, Hamilton J. Motivational interviewing to enhance self-efficacy and promote weight loss in overweight and obese adolescents: a randomized controlled trial. J Pediatr Psychol. 2013 Oct;38(9):944-53. doi: 10.1093/jpepsy/jst023. Epub 2013 May 13. PMID 23671058
- [Background] Flattum C, Friend S, Story M, Neumark-Sztainer D. Evaluation of an individualized counseling approach as part of a multicomponent school-based program to prevent weight-related problems among adolescent girls. J Am Diet Assoc. 2011 Aug;111(8):1218-23. doi: 10.1016/j.jada.2011.05.008. PMID 21802570
- [Derived] Videira-Silva A, de Freitas F, Sardinha LB, Fonseca H. Effect and safety of a physical exercise-based intervention on body composition and cardiometabolic health of adolescents with severe obesity. Secondary analysis from the PAC-MAnO trial. Obes Pillars. 2025 Jun 26;16:100190. doi: 10.1016/j.obpill.2025.100190. eCollection 2025 Dec. PMID 40688482
- [Derived] Videira-Silva A, Santos I, Freaza D, Gameiro M, Sardinha LB, Fonseca H. Dietary content and combined training, but not daily physical activity, are associated with 6-month bone mineral changes in adolescents with obesity: A Secondary analysis of the PAC-MAnO trial. Eur J Pediatr. 2024 Sep;183(9):3969-3978. doi: 10.1007/s00431-024-05659-4. Epub 2024 Jun 27. PMID 38937331
- [Derived] Videira-Silva A, Sardinha LB, Fonseca H. Atherosclerosis Prevention in Adolescents with Obesity: The Role of Moderate-Vigorous Physical Activity. Int J Environ Res Public Health. 2022 Nov 23;19(23):15537. doi: 10.3390/ijerph192315537. PMID 36497620
- [Derived] Videira-Silva A, Hetherington-Rauth M, Sardinha LB, Fonseca H. Combined high-intensity interval training as an obesity-management strategy for adolescents. Eur J Sport Sci. 2023 Jan;23(1):109-120. doi: 10.1080/17461391.2021.1995508. Epub 2021 Nov 12. PMID 34663193
- [Derived] Videira-Silva A, Sardinha L, Fonseca H. Effect of a Physical Activity Consultation in the Management of Adolescent Overweight (the PAC-MAnO project): study rationale, design and methods. BMJ Paediatr Open. 2018 Jul 15;2(1):e000214. doi: 10.1136/bmjpo-2017-000214. eCollection 2018. PMID 30094347